CLINICAL TRIAL: NCT00001449
Title: A Phase I Study of Weekly Gemcitabine in Combination With Infusional Fluorodeoxyuridine and Oral Calcium Leucovorin in Adult Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950197; 95-C-0197
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-09

CONDITIONS: Neoplasms
Keywords: Anti-Cancer Agents; Antimetabolite; Palliation; Pharmacodynamics; Pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — Gemcitabine; Floxuridine; Leucovorin

INTERVENTIONS:
Drug: gemcitabine
Drug: fluorodeoxyuridine
Drug: leucovorin

SUMMARY:
The purpose of this study is to determine the clinical toxicities associated with administering sequential dFdC as a one hour infusion followed by a continuous infusion of FUdR over 24 hours with low dose oral LV weekly for three weeks out of four.

DETAILED DESCRIPTION:
The MTD and biochemically active dose of FUDR as a 24-hour and gemcitabine as a 2-hour infusion will be determined first (Part A); if the biochemically active FUDR dose is less than the MTD, new patients will be entered to determine the maximum tolerated duration of FUDR infusion (Part B).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Diagnostically proven locally advanced, but unresectable primary or recurrent solid tumors or lymphoma or metastatic solid tumors that have failed standard therapy or no such therapy is available.

Objectively measurable disease not required.

No patients with leukemia or primary or metastatic CNS malignancies.

PRIOR/CONCURRENT THERAPY:

Biologic Therapy: Greater than 4 weeks since prior immunotherapy and recovered from all toxic effects.

Chemotherapy: Greater than 4 weeks since prior chemotherapy and recovered from all toxic effects with following exceptions: At least 6 weeks since prior mitomycin C or nitrosourea therapy. At least 3 months since prior suramin therapy.

Endocrine Therapy: Not specified

Radiotherapy: At least 2 weeks since prior radiotherapy (4 weeks if at least 21% of marrow irradiated) and recovered from all toxic effects.

Surgery: Recovered from any prior surgery.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance status: ECOG 0-2

Hematopoietic:

AGC at least 2,000/microL.

Platelet count at least 100,000/microL.

Hepatic: Bilirubin no greater than 2.0 mg/dL.

Renal: Creatinine no greater than 2.0 mg/dL.

OTHER:

No failure of prior gemcitabine therapy.

No concurrent cimetidine (ranitidine and other anti-ulcer agents allowed).

No active infection requiring intravenous antibiotic therapy.

HIV negative.

No other medical contraindication to protocol therapy.

No pregnant or nursing women.

Adequate contraception required of fertile patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1995-09; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Heinemann V, Hertel LW, Grindey GB, Plunkett W. Comparison of the cellular pharmacokinetics and toxicity of 2',2'-difluorodeoxycytidine and 1-beta-D-arabinofuranosylcytosine. Cancer Res. 1988 Jul 15;48(14):4024-31. PMID 3383195
- [Background] Heinemann V, Xu YZ, Chubb S, Sen A, Hertel LW, Grindey GB, Plunkett W. Cellular elimination of 2',2'-difluorodeoxycytidine 5'-triphosphate: a mechanism of self-potentiation. Cancer Res. 1992 Feb 1;52(3):533-9. PMID 1732039
- [Background] Heinemann V, Xu YZ, Chubb S, Sen A, Hertel LW, Grindey GB, Plunkett W. Inhibition of ribonucleotide reduction in CCRF-CEM cells by 2',2'-difluorodeoxycytidine. Mol Pharmacol. 1990 Oct;38(4):567-72. PMID 2233693